CLINICAL TRIAL: NCT02208960
Title: An Integrated Toolkit to Save Newborn Lives and Brains in Kenya
Brief Title: Newborn Kit to Save Lives and Brains in Kenya
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Grand Challenges Canada (Other); March of Dimes (Other); Aga Khan University (Other)
Responsible Party: Principal Investigator, Shaun Morris, Associate Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1000044053
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Neurodevelopment; Neonatal Mortality
Keywords: Neurodevelopment; Neonatal kit; Kenya; Cluster Randomized Controlled Trial; Chlorhexidine; ThermoSpot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Neonatal Kit (Experimental): Mothers in the neonatal kit clusters will receive a neonatal kit and training on how to use the kit components during their third trimester of pregnancy. The kit will contain a clean birth kit to be used at the time of delivery either at home or in a facility, 4% chlorhexidine (CHX) lotion, sunflower oil emollient, ThermoSpot, a Mylar infant sleeve, and a reusable, non-electric, heating device. Community Health Workers will be equipped with a hand-held battery operated scale to identify low birth weight newborns.
  Interventions: Device: Neonatal Kit
- Neonatal Stimulation (Experimental): During home visits in the 3rd trimester, mothers in the neonatal stimulation clusters will be taught 3 core messages pertaining to neonatal stimulation. First, mothers will be taught how to make eye contact and talk to their child. This type of interaction encourages social inclusion, attachment, and development of social-communication skills. Second, mothers will be taught techniques to foster responsive feeding and caregiving. Finally, mothers will be encouraged to sing songs and nursery rhymes, including those with gentle touch in order to support the development of communication skills, and introduce a tactile component to caregiving. These messages will be reiterated at subsequent home visits by the CHW after the baby is born.
  Interventions: Behavioral: Neonatal Stimulation
- Neonatal Kit and Neonatal Stimulation (Experimental): Participants in this arm of the study will receive both a neonatal kit (described in Arm 1) and neonatal stimulation (described in Arm 2).
  Interventions: Device: Neonatal Kit; Behavioral: Neonatal Stimulation
- Control (Standard Care) (No Intervention): In control clusters, CHWs will visit the home according to the regular schedule (same as in the intervention clusters) and deliver the standard CHW post-natal care that consists of talking to mothers about:
  * Exclusive breastfeeding and proper nutrition for both the mother and the baby.
  * Ensuring warmth to the baby.
  * Full immunization and growth monitoring of newborn.
  * Hygiene and sanitation practices.
  * Family Planning and promote the proper use of Insecticides Treated Nets.
  * Identifying any danger sign/complication for both mothers and new-borns and refer for prompt treatment (within 24 hours) for management and treatment.
  * Promoting the use of services such as birth registration.
  * Giving advice on proper care of the umbilical cord.

INTERVENTIONS:
Device: Neonatal Kit — Contents of the neonatal kit:
  1. Clean birth kit: sterile blade, a clean plastic square, plastic gloves, hand soap, and cord ties/clamp.
  2. 4% Chlorhexidine (CHX) lotion (15 mL) and a bag of cotton balls.
  3. Sunflower oil emollient (50 mL)
  4. ThermoSpot
  5. Mylar infant sleeve
  6. Click to heat warmer (http://www.heatinaclick.ca/products/pocket_size.html) in a fitted cloth pouch.
  7. Handheld battery-operated scale with suspended cloth sling. The scale will not be included with the kit but rather one will be issued to each Community Health Worker.
  Arms: Neonatal Kit; Neonatal Kit and Neonatal Stimulation
Behavioral: Neonatal Stimulation — A sub-set of children in the study will receive a neonatal stimulation program either on its own or in combination with the neonatal kit described above. The stimulation program will focus on teaching three key messages to enhance the caregivers' current caregiving practices, and each message is to be integrated into daily activities (e.g. during feeding, bathing, bedtime routines). By integrating the delivery of the interventions into the caregivers' daily routine, no additional time inconvenience will be added to their schedules. The key messages include:
  1. Eye contact and talking to children
  2. Responsive feeding and caregiving
  3. Singing songs, including those with gentle touch
  Arms: Neonatal Kit and Neonatal Stimulation; Neonatal Stimulation

SUMMARY:
Each year, more than 3 million neonatal deaths occur worldwide and greater than 200 million children under the age of 5, almost all in low- and middle-income countries, are not fulfilling their developmental potential. The development of the growing brain can be affected through multiple mechanisms including the same insults that are major causes of mortality, namely hypothermia and infection. The first month of life is a crucial period in neurodevelopment (ND). In this study, the investigators propose the home-based use of an integrated evidence-based toolkit to improve health status, reduce the incidence of neonatal insults that may affect brain development, decrease neonatal mortality rate (NMR), and provide early identification of danger signs. The investigators hypothesize that use of the neonatal toolkit will result in an improvement of at least one standard deviation in neurodevelopment as measured at 12 months of age by the Protocol for Child Monitoring Infant and Toddler (PCM-IT) version.

DETAILED DESCRIPTION:
Each year there are over 3 million global neonatal deaths. While significant progress has been made on overall under 5 mortality over the past decade, minimal progress has been made in reducing neonatal deaths and these now represent about 40% of all deaths in children under the age of 5. The majority of neonatal deaths occur in rural areas of developing countries and approximately two thirds are due to infection and complications relating to low birth weight (LBW) and prematurity. Additionally, more than 200 million children under 5 years old, almost all in low- and middle-income countries (LMIC), are not fulfilling their developmental potential. To date, most neonatal intervention trials in LMIC have focused on reducing mortality and little research has been performed on the consequences of severe but non-fatal neonatal insults on neurodevelopment (ND). Subsequently, little is known about interventions that may reduce the risk of long-term neurocognitive sequelae.

The first month of life is a critical period in ND in which there is significant neurogenesis, synaptogenesis, and myelination. Stimulation of the infant's brain during this period may have significant downstream positive effects. Development of the growing brain can be affected through multiple mechanisms including the same insults that are major causes of mortality, namely hypothermia and infection. Reducing the incidence of these insults during this period may not only save lives but also save brains and improve ND outcomes.

ELIGIBILITY:
Inclusion Criteria:

i. All pregnant women in parts of study clusters covered by CHW program and their home- or facility-born live newborns.

ii. Mothers intending to maintain residence in study area for first 12 months of newborn's life.

Exclusion Criteria:

i. Failure to provide consent to enroll in study (intervention or control clusters).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2294 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Neurodevelopment as measured by the Protocol for Child Monitoring - Infant and Toddler version assessment | 12 months of age
  The Protocol for Child Monitoring - Infant and Toddler (PCM-IT) version was designed in Kenya to assess neurodevelopment in resource-limited settings.

SECONDARY OUTCOMES:
Neonatal mortality | Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life
  Death from any cause within the first 28 days of life
Incidence of omphalitis | Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life
  Incidence of omphalitis where omphalitis is defined as:
  1. None (no redness or swelling)
  2. Mild (inflammation limited to the cord stump)
  3. Moderate (inflammation extending less than 2cm to the skin at the base of the cord stump)
  4. Severe (inflammation extending more than 2cm from the cord stump)
Incidence of severe infection | Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life
  Defined as:
  Convulsions OR fast breathing (60 breaths per minute or more) OR severe chest indrawing OR movement only when stimulated or no movement at all OR not feeding at all for at least 12 hours.
Cases of hypothermia identified | Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life
  Defined using ThermoSpot as:
  1. Moderate hypothermia: pale green and red face (35ºC to 36ºC)
  2. Severe hypothermia: black face (<35ºC)
Cases of hyperthermia identified | Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life
  Defined using ThermoSpot as:
  Hyperthermia: blue face (>39ºC)
Number of LBW babies identified | Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life
  LBW defined as: <2500 grams at first weighing
Health facility use | Day 1 (or as soon as possible after notification of birth), 3, 7, 14, and 28 of life

CONTACTS AND LOCATIONS:
Overall Officials: Shaun K Morris, MD, MPH, Principal Investigator — The Hospital for Sick Children; Robert Armstrong, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Nairobi, Kenya

REFERENCES:
- [Background] Abubakar A, Holding P, van Baar A, Newton CR, van de Vijver FJ. Monitoring psychomotor development in a resource-limited setting: an evaluation of the Kilifi Developmental Inventory. Ann Trop Paediatr. 2008 Sep;28(3):217-26. doi: 10.1179/146532808X335679. PMID 18727851
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Lawn JE, Kinney MV, Black RE, Pitt C, Cousens S, Kerber K, Corbett E, Moran AC, Morrissey CS, Oestergaard MZ. Newborn survival: a multi-country analysis of a decade of change. Health Policy Plan. 2012 Jul;27 Suppl 3:iii6-28. doi: 10.1093/heapol/czs053. PMID 22692417
- [Background] Arifeen SE, Mullany LC, Shah R, Mannan I, Rahman SM, Talukder MR, Begum N, Al-Kabir A, Darmstadt GL, Santosham M, Black RE, Baqui AH. The effect of cord cleansing with chlorhexidine on neonatal mortality in rural Bangladesh: a community-based, cluster-randomised trial. Lancet. 2012 Mar 17;379(9820):1022-8. doi: 10.1016/S0140-6736(11)61848-5. Epub 2012 Feb 8. PMID 22322124
- [Background] Darmstadt GL, Saha SK, Ahmed AS, Ahmed S, Chowdhury MA, Law PA, Rosenberg RE, Black RE, Santosham M. Effect of skin barrier therapy on neonatal mortality rates in preterm infants in Bangladesh: a randomized, controlled, clinical trial. Pediatrics. 2008 Mar;121(3):522-9. doi: 10.1542/peds.2007-0213. PMID 18310201
- [Background] Mullany LC, Darmstadt GL, Khatry SK, Katz J, LeClerq SC, Shrestha S, Adhikari R, Tielsch JM. Topical applications of chlorhexidine to the umbilical cord for prevention of omphalitis and neonatal mortality in southern Nepal: a community-based, cluster-randomised trial. Lancet. 2006 Mar 18;367(9514):910-8. doi: 10.1016/S0140-6736(06)68381-5. PMID 16546539
- [Background] Mullany LC, El Arifeen S, Winch PJ, Shah R, Mannan I, Rahman SM, Rahman MR, Darmstadt GL, Ahmed S, Santosham M, Black RE, Baqui AH. Impact of 4.0% chlorhexidine cleansing of the umbilical cord on mortality and omphalitis among newborns of Sylhet, Bangladesh: design of a community-based cluster randomized trial. BMC Pediatr. 2009 Oct 21;9:67. doi: 10.1186/1471-2431-9-67. PMID 19845951
- [Background] Khan A, Kinney MV, Hazir T, Hafeez A, Wall SN, Ali N, Lawn JE, Badar A, Khan AA, Uzma Q, Bhutta ZA; Pakistan Newborn Change and Future Analysis Group. Newborn survival in Pakistan: a decade of change and future implications. Health Policy Plan. 2012 Jul;27 Suppl 3:iii72-87. doi: 10.1093/heapol/czs047. PMID 22692418
- [Derived] Pell LG, Bassani DG, Nyaga L, Njagi I, Wanjiku C, Thiruchselvam T, Macharia W, Minhas RS, Kitsao-Wekulo P, Lakhani A, Bhutta ZA, Armstrong R, Morris SK. Effect of provision of an integrated neonatal survival kit and early cognitive stimulation package by community health workers on developmental outcomes of infants in Kwale County, Kenya: study protocol for a cluster randomized trial. BMC Pregnancy Childbirth. 2016 Sep 8;16(1):265. doi: 10.1186/s12884-016-1042-5. PMID 27608978